CLINICAL TRIAL: NCT00379262
Title: Randomized Trial to Evaluate Therapeutic Gain by Changing Chemoradiotherapy From Concurrent-adjuvant to Induction-concurrent Sequence, and Radiotherapy From Conventional to Accelerated Fractionation for Advanced Nasopharyngeal Carcinoma
Brief Title: Therapeutic Gain by Induction-concurrent Chemoradiotherapy and/or Accelerated Fractionation for Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hong Kong Nasopharyngeal Cancer Study Group Limited (Other)
Collaborators: The Hong Kong Anti-Cancer Society (Other); hong Kong Cancer Fund (Unknown)
Responsible Party: Principal Investigator, Dr. ANNE W M LEE, Consultant, Dept of Clinical Oncology, PYNEH, Hong Kong Nasopharyngeal Cancer Study Group Limited
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NPC-0501 Trial
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Chemoradiotherapy; Accelerated Fractionation
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Capecitabine; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1A (Experimental): Concurrent-Adjuvant CRT using P-PF regimen and conventional fractionation radiotherapy
  Interventions: Drug: Adjuvant chemotherapy using PF (5-Fluorouracil )
- 1B (Experimental): Concurrent-Adjuvant CRT using P-PF regimen and accelerated fractionation radiotherapy
  Interventions: Drug: Adjuvant chemotherapy using PF (5-Fluorouracil )
- 2A (Experimental): Induction-Concurrent CRT using PF-P regimen and conventional fractionation radiotherapy
  Interventions: Drug: Induction chemotherapy using PF (5-Fluorouracil)
- 2B (Experimental): Induction-Concurrent CRT using PF-P regimen and accelerated fractionation radiotherapy
  Interventions: Drug: Induction chemotherapy using PF (5-Fluorouracil)
- 3A (Experimental): Induction-Concurrent CRT using PX-P regimen and conventional fractionation radiotherapy
  Interventions: Drug: Capecitabine
- 3B (Experimental): Induction-Concurrent CRT using PX-P regimen and accelerated fractionation radiotherapy
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Dose:1000 mg/m2, BD, Day 1-Day 14 Interval: 21 days Cycles: 3 cycles
  Other Names: Xeloda
  Arms: 3A; 3B
Drug: Adjuvant chemotherapy using PF (5-Fluorouracil ) — Cisplatin 80 mg/m2 IV + 5-Fluorouracil 1000 mg/m2/day IV infusion for 96 hr every 28 days for 3 cycles
  Arms: 1A; 1B
Drug: Induction chemotherapy using PF (5-Fluorouracil) — Cisplatin 100 mg/m2 IV + 5-Fluorouracil 1000 mg/m2/day IV infusion for 120 hr every 21 days for 3 cycles
  Arms: 2A; 2B

SUMMARY:
The objectives of this clinical study are threefold:

1. To compare the benefits in cancer control and survival obtained from adding induction-concurrent chemotherapy to radiation with those from adding concurrent-adjuvant chemotherapy to radiation.
2. To test whether replacing fluorouracil with Xeloda in combining with cisplatin in the chemotherapy plan will maintain or improve further the chemotherapy benefits while reducing the duration of hospital stay.
3. To see if accelerated fractionation radiotherapy can improve the outcome of patients as compared with conventional fractionation radiotherapy.

DETAILED DESCRIPTION:
1. primary objectives include

   1. comparing induction chemotherapy with Cisplatin + 5-Fluorouracil versus adjuvant chemotherapy with Cisplatin + 5-Fluorouracil(PF-Pvs P-PF)
   2. comparing induction chemotherapy with Cisplatin + Capecitabine versus adjuvant chemotherapy with Cisplatin + 5-Fluorouracil(PX-P vs P-PF)
   3. comparing accelerated fractionation versus conventional fractionation (AF vs CF)radiotherapy.
2. secondary objectives include

   1. comparing induction chemotherapy with Cisplatin + Capecitabine versus induction chemotherapy with Cisplatin + 5-Fluorouracil(PX-P vs PX-P)
   2. Comparing concurrent-adjuvant (CA) versus induction-concurrent (IC) chemotherapy sequence.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven nasopharyngeal carcinoma for primary treatment with radical intent
* non-keratinizing or undifferentiated type
* stage III-IVB (by AJCC/UICC 6th edition)
* ECOG Performance status less or equal to 2
* Marrow: WBC >= 4 and platelet >=100
* Renal: creatinine clearance >=60
* Informed consent

Exclusion Criteria:

* Primary treatment with palliative intent
* WHO type I squamous cell carcinoma or adenocarcinoma
* Evidence of distant metastases
* Patient is pregnant or lactating
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer or other cancer for which the patient has been disease-free for 5 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 803 (Actual)
Dates: Start 2006-09; Primary Completion 2017-05 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival, defined as the time to treatment failure at any site or death due to any cause, at 5-year. | 5 years
Overall Survival, defined as the time to death due to any cause, at 5-year. | 5 years

SECONDARY OUTCOMES:
overall Failure-Free Rate, defined as time to failure at any site) | 5 years
Loco-regional Failure-Free Rate, defined as time to local or nodal failure) | 5 years
Distant Failure-Free Rate, defined as time to distant failure) | 5 years
Incidence of chemotherapy toxicity and acute RT toxicity grade > 3 | treatment
Time to late toxicity (From the date of randomization to the earliest date of late toxicity grade > 3) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Anne W.M. Lee, F.R.C.R., Principal Investigator — Department of Clinical Oncology, Pamela Youde Nethersole Eastern Hospital, Hong Kong; Roger K.C. Ngan, F.R.C.R, Principal Investigator — Department of Clinical Oncology, Quen Elizabeth Hospital, Hong Kong
Locations (7):
- China (7):
  - Cancer Center, Sun Yat Sen University, Guangzhou
  - Department of Clinical Oncology, Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong
  - Department of Clinical Oncology, Princess Margaret Hospital, Hong Kong
  - Department of Clinical Oncology, Queen Elizabeth Hospital, Hong Kong
  - Department of Clinical Oncology, Queen Mary Hospital, Hong Kong
  - Department of Clinical Oncology, Tuen Mun Hospital, Hong Kong

REFERENCES:
- [Background] Al-Sarraf M, LeBlanc M, Giri PG, Fu KK, Cooper J, Vuong T, Forastiere AA, Adams G, Sakr WA, Schuller DE, Ensley JF. Chemoradiotherapy versus radiotherapy in patients with advanced nasopharyngeal cancer: phase III randomized Intergroup study 0099. J Clin Oncol. 1998 Apr;16(4):1310-7. doi: 10.1200/JCO.1998.16.4.1310. PMID 9552031
- [Background] Lee AW, Lau WH, Tung SY, Chua DT, Chappell R, Xu L, Siu L, Sze WM, Leung TW, Sham JS, Ngan RK, Law SC, Yau TK, Au JS, O'Sullivan B, Pang ES, O SK, Au GK, Lau JT; Hong Kong Nasopharyngeal Cancer Study Group. Preliminary results of a randomized study on therapeutic gain by concurrent chemotherapy for regionally-advanced nasopharyngeal carcinoma: NPC-9901 Trial by the Hong Kong Nasopharyngeal Cancer Study Group. J Clin Oncol. 2005 Oct 1;23(28):6966-75. doi: 10.1200/JCO.2004.00.7542. PMID 16192584
- [Background] Lee N, Xia P, Quivey JM, Sultanem K, Poon I, Akazawa C, Akazawa P, Weinberg V, Fu KK. Intensity-modulated radiotherapy in the treatment of nasopharyngeal carcinoma: an update of the UCSF experience. Int J Radiat Oncol Biol Phys. 2002 May 1;53(1):12-22. doi: 10.1016/s0360-3016(02)02724-4. PMID 12007936
- [Background] Le QT, Tate D, Koong A, Gibbs IC, Chang SD, Adler JR, Pinto HA, Terris DJ, Fee WE, Goffinet DR. Improved local control with stereotactic radiosurgical boost in patients with nasopharyngeal carcinoma. Int J Radiat Oncol Biol Phys. 2003 Jul 15;56(4):1046-54. doi: 10.1016/s0360-3016(03)00117-2. PMID 12829140
- [Background] Baujat B, Audry H, Bourhis J, Chan AT, Onat H, Chua DT, Kwong DL, Al-Sarraf M, Chi KH, Hareyama M, Leung SF, Thephamongkhol K, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy in locally advanced nasopharyngeal carcinoma: an individual patient data meta-analysis of eight randomized trials and 1753 patients. Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):47-56. doi: 10.1016/j.ijrobp.2005.06.037. PMID 16377415
- [Background] Hoff PM, Ansari R, Batist G, Cox J, Kocha W, Kuperminc M, Maroun J, Walde D, Weaver C, Harrison E, Burger HU, Osterwalder B, Wong AO, Wong R. Comparison of oral capecitabine versus intravenous fluorouracil plus leucovorin as first-line treatment in 605 patients with metastatic colorectal cancer: results of a randomized phase III study. J Clin Oncol. 2001 Apr 15;19(8):2282-92. doi: 10.1200/JCO.2001.19.8.2282. PMID 11304782
- [Background] Twelves C, Boyer M, Findlay M, Cassidy J, Weitzel C, Barker C, Osterwalder B, Jamieson C, Hieke K; Xeloda Colorectal Cancer Study Group. Capecitabine (Xeloda) improves medical resource use compared with 5-fluorouracil plus leucovorin in a phase III trial conducted in patients with advanced colorectal carcinoma. Eur J Cancer. 2001 Mar;37(5):597-604. doi: 10.1016/s0959-8049(00)00444-5. PMID 11290435
- [Background] Chua DT, Sham JS, Au GK. A phase II study of capecitabine in patients with recurrent and metastatic nasopharyngeal carcinoma pretreated with platinum-based chemotherapy. Oral Oncol. 2003 Jun;39(4):361-6. doi: 10.1016/s1368-8375(02)00120-3. PMID 12676255
- [Background] Greene FL, et al. AJCC Cancer Staging Handbook from the AJCC cancer staging manual, 6th ed. New York: Springer, 2002.
- [Background] Lee AW, Tung SY, Chan AT, Chappell R, Fu YT, Lu TX, Tan T, Chua DT, O'sullivan B, Xu SL, Pang ES, Sze WM, Leung TW, Kwan WH, Chan PT, Liu XF, Tan EH, Sham JS, Siu L, Lau WH. Preliminary results of a randomized study (NPC-9902 Trial) on therapeutic gain by concurrent chemotherapy and/or accelerated fractionation for locally advanced nasopharyngeal carcinoma. Int J Radiat Oncol Biol Phys. 2006 Sep 1;66(1):142-51. doi: 10.1016/j.ijrobp.2006.03.054. PMID 16904519
- [Background] Freedman J, Furberg, C, DeMets D. Fundamentals of clinical trials. Springer-Verlag, NY, 1998.